CLINICAL TRIAL: NCT02747914
Title: Repetitive Transcranial Magnetic Stimulation Boosted Exercise Therapy for Lower Limb Spasticity in Multiple Sclerosis Patients
Brief Title: Repetitive Transcranial Magnetic Stimulation for Lower Limb Spasticity in Multiple Sclerosis Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK-5
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial magnetic stimulation therapy (Experimental): Group of patients treated with rTMS low than 5Hz
  Interventions: Device: Transcranial magnetic stimulation
- Conventional exercise treatment (Active Comparator): Group of patients treated with conventional exercise
  Interventions: Other: Conventional exercise

INTERVENTIONS:
Device: Transcranial magnetic stimulation — TMS 1Hz under the motor zone of cortex.
  Arms: Transcranial magnetic stimulation therapy
Other: Conventional exercise — Exercise will be administrated in a conventional way.
  Arms: Conventional exercise treatment

SUMMARY:
Leg spasticity is common problem encountered with a large proportion of patients suffering with multiple sclerosis (MS) with an increasing severity as the disease progresses. It mostly affects the antigravity muscles that significantly complicates transfer, increases fatigue and makes walking more difficult. Hence, leg spasticity often interferes with patients' mobility and significantly influences their quality of life. A great number of multidisciplinary rehabilitation studies has shown a significant effect of numerous specific functional changes in patients with secondary (SP) and primary progressive (PP) MS but there are no reviews related to spasticity. The positive therapeutic effect of modulating Transcranial Magnetic Stimulation ( TMS) methods on spasticity is shown in only two studies, in patients with relapse remitting clinical form in the remission phase of the disease. The effect of TMS on clinical measures of lower limb spasticity, functional inability and the quality of life in patients with SPMS and PPMS will be examined in this study. The objective to this study are to to explore whether rTMS boosted exercise therapy (ET) treatment can bring more improvement in lower limb spasticity than ET treatment alone in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical form of SPMS and PPMS (established on the basis of the revised McDonald criteria)
* EDDS score 2-6.5
* lower limb spasticity caused by MS
* 18 years ≥age of the patient ≤ 65. years

Exclusion Criteria:

* clinical worsening of the disease over the past 30 days,
* the presence of pregnancy, dementia, alcoholism, history of loss of consciousness, epilepsy, metal objects in the head, pacemakers and other electronic devices in the body at a distance of 20cm from the top of the patients head, serious associate diseases (malignancy, heart disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
muscle tone measured by Modified Ashworth Scale (MAS) | 3 weeks

SECONDARY OUTCOMES:
impact of leg spasticity on daily activities measured by Multiple Sclerosis Spasticity Scale 88 (MSSS-88) | 3 weeks
Activities of daily living measured by Barthel Index | 3 weeks
Walking mobility measured by Timed 25 Foot Walk test | 3 weeks
Quality of life measured by Multiple Sclerosis Quality of Life 54 (MSQoL54). | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia